CLINICAL TRIAL: NCT06246903
Title: INTER-PATHOLOGIST READER STUDY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Orlucent, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SFI006
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Nevi, Dysplastic
MeSH Terms: conditions — Dysplastic Nevus Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspicious nevus/nevi

SUMMARY:
This is a post study histology analysis from previously obtained pathology slides.

DETAILED DESCRIPTION:
This is a post study histology analysis. Pathologists will use digital histology slide scans of suspicious nevus/nevi obtained from previously conducted studies to provide histopathology gradations of histological features as outlined in the Orlucent histology atlas (LBL0713 Histopathology Atlas for Grading of Dysplastic Nevi and DEF0713-1 Histopathology Definitions for LBL0713).

ELIGIBILITY:
Inclusion Criteria:

1. Histology scans must have been obtained from previous consented subjects that allows post study ad hoc analyses.
2. Histology scans must be available from the data collected from the Orlucent OMS002, SFI001 or SFI003 Studies and are of good quality.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previous consented subject's scans from the Orlucent OMS002, SFI001 or SFI003 Studies and
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Study Success | 8 months
  This is a data collection study. Study success is considered when the interpathology agreement is improved when compared to the agreement identified in Elmore et al. [5]. [(classes/agreement): class I (eg, nevus or mild atypia) / 92% (95% confidence interval 90% to 94); class II (eg, moderate atypia) / 25% (22% to 28%); III (eg, severe atypia or melanoma in situ) / 40% (37% to 44%); IV (eg, pathologic stage T1a (pT1a) early invasive melanoma) / 43% (39% to 46%); and V (eg, ≥pT1b invasive melanoma) / 72% (69% to 75%).]

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Shachaf, PhD, Study Director — Founder and President
Locations (1):
- University of Utah Hospital, Pathology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided